CLINICAL TRIAL: NCT01227278
Title: A Phase 2a, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of MEDI-563 in Subjects With Moderate-to-severe Chronic Obstructive Pulmonary Disease and Sputum Eosinophilia
Brief Title: A Study to Evaluate the Effectiveness of MEDI-563 in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP196; 2010-020127-52 (EudraCT Number)
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Benralizumab; MEDI-563; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to benralizumab (MEDI-563) injection subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks for the next 5 doses (Day 1, 29, 57, 113, 169, 225, 281 and 337).
  Interventions: Other: Placebo
- Benralizumab 100 mg (Experimental): Benralizumab (MEDI-563) 100 mg injection subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks for the next 5 doses (Day 1, 29, 57, 113, 169, 225, 281 and 337).
  Interventions: Biological: Benralizumab 100 mg

INTERVENTIONS:
Other: Placebo — Placebo matched to benralizumab (MEDI-563) injection subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks for the next 5 doses (Day 1, 29, 57, 113, 169, 225, 281 and 337).
  Arms: Placebo
Biological: Benralizumab 100 mg — Benralizumab (MEDI-563) 100 mg injection subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks for the next 5 doses (Day 1, 29, 57, 113, 169, 225, 281 and 337).
  Other Names: MEDI-563
  Arms: Benralizumab 100 mg

SUMMARY:
To evaluate the effect of the drug in moderate to severe Chronic Obstructive Pulmonary Disease (COPD) in Adults.

DETAILED DESCRIPTION:
To evaluate the effect of multiple subcutaneous (SC) doses of benralizumab (MEDI 563) on the rate of moderate-to-severe annualized incidence rate of moderate or severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD) in adult subjects with moderate-to-severe COPD who exhibit eosinophilia (greater than or equal to [>=] 3.0 percent [%] sputum eosinophilia in the previous 12 months or at Screening) in sputum compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 40-85 years at the time of Screening
* Written informed consent obtained from the subject prior to performing any protocol related procedures
* Documented history of 1 or more Annualized Incidence Rate of Moderate or Severe Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
* Current smoker or ex-smoker with a tobacco history of greater than or equal to (>=) 10 pack-years
* Adequate contraception from screening through end of trial
* Able to read and write.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Pregnant, breastfeeding, or lactating women
* Known history of allergy or reaction to any component of the investigational product formulation
* History of anaphylaxis to any other biologic therapy
* Donation or transfusion of blood, plasma or platelets within the past 3 months prior to Screening
* Other significant pulmonary disease which in the opinion of the investigator or medical monitor, might compromise the interpretation of the study
* Fever greater than (>) 37.0 degree Centigrade (98.6 degree Fahrenheit) at Screening
* Receipt of any novel investigational medicinal product within 3 months before the first dose of investigational product in this study and through the end of the study
* Seropositive for hepatitis A, hepatitis B surface antigen, hepatitis C, or human immunodeficiency virus 1or 2 (HIV-1 or HIV 2)
* History of alcohol or drug abuse within the past year that required treatment that the investigator felt or medical monitor felt would compromise the study data interpretation
* Past or current malignancy within the past 5 years except adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma in situ treated with apparent success more than 1 year prior to Screening
* Subjects participating in, or scheduled for, an intensive COPD rehabilitation program (subjects who are in the maintenance phase of a rehabilitation program are eligible to take part)
* Current diagnosis of asthma according to Global Initiative for Asthma guidelines
* Previous treatment with MEDI-563.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene van der Merwe, MBChB, Study Director — MedImmune Ltd
Locations (31):
- United States (9):
  - Research Site, Los Angeles, California
  - Research Site, Marietta, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Brooklyn, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Greenville, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Tyler, Texas
  - Research Site, Richmond, Virginia
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Denmark (4):
  - Research Site, Århus C
  - Research Site, Hellerup
  - Research Site, København NV
  - Research Site, Odense C
- Germany (2):
  - Research Site, Frankfurt
  - Research Site, Mainz
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Lleida
  - Research Site, Málaga
  - Research Site, Oviedo
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Leicester
  - Research Site, Manchester

REFERENCES:
- [Derived] Sridhar S, Liu H, Pham TH, Damera G, Newbold P. Modulation of blood inflammatory markers by benralizumab in patients with eosinophilic airway diseases. Respir Res. 2019 Jan 18;20(1):14. doi: 10.1186/s12931-018-0968-8. PMID 30658649
- [Derived] Brightling CE, Bleecker ER, Panettieri RA Jr, Bafadhel M, She D, Ward CK, Xu X, Birrell C, van der Merwe R. Benralizumab for chronic obstructive pulmonary disease and sputum eosinophilia: a randomised, double-blind, placebo-controlled, phase 2a study. Lancet Respir Med. 2014 Nov;2(11):891-901. doi: 10.1016/S2213-2600(14)70187-0. Epub 2014 Sep 7. PMID 25208464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 421 participants were screened and 101 participants were randomized into the study.
Groups:
- Benralizumab 100 mg: Benralizumab (MEDI-563) 100 milligram (mg) injection subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks for the next 5 doses (Day 1, 29, 57, 113, 169, 225, 281 and 337).
Period: Overall Study
Arm/Group | Placebo | Benralizumab 100 mg
Started | 50 | 51
Completed | 45 | 43
Not Completed | 5 | 8
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Death | 0 | 2
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Benralizumab 100 mg | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.5) | 62.9 (8.2) | 63.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 29 | 35 | 64

OUTCOME MEASURES:

1. Primary Outcome: Annualized Incidence Rate of Moderate or Severe Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: An AECOPD is defined as worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days. Annualized Incidence Rate of Moderate or Severe AECOPD was assessed based on AECOPD data up to Day 393 (Rate = total number of moderate or severe AECOPD in each group/total person-year follow-up in each group). The severity of an exacerbation of COPD is defined as: a) Mild exacerbations, which require treatment with an increase in usual therapy, example (eg), increase use of short acting bronchodilators, b) Moderate exacerbations which require treatment with systemic corticosteroids, and or antibiotics and c) Severe exacerbations which require hospitalization.
Time Frame: Day 1 up to 393
Population: The per protocol (PP) population included all participants who had no major protocol violations, received at least 6 of the 8 total doses of investigational product, and completed the study through Day 393.
Measure: Number (95% Confidence Interval); unit: AECOPD events/person-year
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
AECOPD events/person-year | 0.92 [0.67 to 1.25] | 0.95 [0.68 to 1.29]
Statistical Analysis 1: Comparison: Placebo vs Benralizumab 100 mg; Test type: Superiority or Other; p = 0.941, Van Elteren Test; Day 1 to 393: Van Elteren test was used to compare the two arms; Rate ratio = 1.03, 95% CI 2-sided [0.67 to 1.58] — 95 percent (%) confidence interval (CI) for rate ratio was based on normal approximation assuming rate with Poisson distribution

2. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to Day 561 that were absent before treatment or that worsened relative to pre-treatment state. TEAEs reported below included both SAEs and non-serious AEs.
Time Frame: Day 1 up to 561
Population: The safety population included all participants who received at least one dose of investigational drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 50 | 51
participants
  TEAEs | 41 | 45
  TESAEs | 9 | 14

3. Secondary Outcome: Number of Participants Hospitalized Due to Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: An AECOPD is defined as worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days.
Time Frame: Day 1 up to 393
Population: The PP population included all participants who had no major protocol violations, received at least 6 of the 8 total doses of investigational product, and completed the study through Day 393.
Measure: Number; unit: participants
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
participants | 5 | 2

4. Secondary Outcome: Percentage of Participants Hospitalized Due to Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: as for outcome 3
Time Frame: Day 1 up to 393
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
percentage of participants | 11.9 | 5.0

5. Secondary Outcome: Annual Incidence Rate of Hospitalization Due to Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: An AECOPD is defined as worsening of two or more major symptoms or one major and one minor symptom for two or more consecutive days. Annualized Incidence Rate of hospitalization due to AECOPD was calculated as Rate = total number of hospitalizations/ total person years.
Time Frame: Day 1 up to 393
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: hospitalizations/person-year
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
hospitalizations/person-year | 0.11 [0.05 to 0.26] | 0.05 [0.01 to 0.18]

6. Secondary Outcome: Change From Baseline in COPD-Specific Saint George's Respiratory Questionnaire (SGRQ-C) Total and Domain Scores at Day 393
Description: The SGRQ is a health related quality of life questionnaire consisting of 40 items in three domains: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response has a unique empirically derived weight where lowest possible weight is zero and the highest is 100. The total score and domain score are derived from the relevant items and converted to a score of 0 to 100 with a higher score indicating poorer health status.
Time Frame: Baseline, Day 393
Population: The PP population included all participants who had no major protocol violations, received at least 6 of the 8 total doses of investigational product, and completed the study through Day 393. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
units on scale
  Baseline: Total Score (n=42, 40) | 48.04 (19.14) | 51.75 (20.45)
  Change at Day 393: Total Score (n=42, 37) | -4.43 (11.71) | -5.51 (16.64)
  Baseline: Symptoms (n=42, 40) | 64.59 (24.38) | 67.18 (21.47)
  Change at Day 393: Symptoms (n=42, 37) | -3.19 (17.44) | -9.02 (21.27)
  Baseline: Activity (n=42, 40) | 58.85 (23.22) | 61.45 (25.53)
  Change at Day 393: Activity (n=42, 37) | -5.65 (14.85) | -4.37 (24.89)
  Baseline: Impact (n=42, 40) | 35.94 (18.95) | 40.69 (22.49)
  Change at Day 393: Impact (n=42, 37) | -4.16 (14.62) | -4.95 (16.97)

7. Secondary Outcome: Percentage of Participants With Improvement in COPD-Specific Saint George's Respiratory Questionnaire (SGRQ-C) Total Score
Description: SGRQ is a health related quality of life questionnaire consisting of 40 items in three domains: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Each question's response has a unique empirically derived weight where lowest possible weight is zero and the highest is 100. The total score and domain score were derived from the relevant items and converted to a score of 0 to 100 with a higher score indicating poorer health status. Percentage of participants with 4-point, 8-point and 12-point change from baseline in SGRQ-C total score were observed.
Time Frame: Day 393
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
percentage of participants
  Day 393, Total: 4-point change (n=42, 37) | 59.5 | 54.1
  Day 393: 8-point change (n=42, 37) | 38.1 | 40.5
  Day 393, Total: 12-point change (n=42, 37) | 21.4 | 24.3

8. Secondary Outcome: Change From Baseline in Chronic Respiratory Questionnaire Self-Administered Standardized Format (CRQ-SAS) Domain Scores at Day 393
Description: The CRQ-SAS is a self-administered questionnaire which consist of 20 items across four domains: dyspnea (5 items), fatigue (4 items), emotional function (7 items), and mastery (4 items). Participants rated their experience on a 7-point scale in response to each item ranging from 1 (maximum impairment) to 7 (no impairment). Individual items were equally weighted, and domain scores were calculated as the mean of all items within each domain; domain score range: 1 (maximum impairment) to 7 (no impairment).
Time Frame: Baseline, Day 393
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
units on scale
  Baseline: Dyspnea (n=42, 40) | 4.97 (1.45) | 4.74 (1.32)
  Change at Day 393: Dyspnea (n=42, 37) | -0.08 (1.29) | 0.09 (1.00)
  Baseline: Fatigue (n=42, 40) | 4.38 (1.26) | 3.96 (1.40)
  Change at Day 393: Fatigue (n=42, 37) | 0.11 (0.94) | 0.11 (1.15)
  Baseline: Emotional function (n=42, 40) | 4.84 (1.24) | 4.72 (1.17)
  Change at Day 393: Emotional function (n=42, 37) | 0.18 (0.98) | 0.08 (1.18)
  Baseline: Mastery (n=42, 40) | 4.89 (1.50) | 4.67 (1.40)
  Change at Day 393: Mastery (n=42, 37) | 0.24 (1.12) | 0.28 (1.24)

9. Secondary Outcome: Percentage of Participants With a 0.5-Point Improvement in Chronic Respiratory Questionnaire Self-administered Standardized Format (CRQ-SAS) Domain Scores at Day 393
Description: The CRQ-SAS is a self-administered questionnaire which consist of 20 items across four domains: dyspnea (5 items), fatigue (4 items), emotional function (7 items), and mastery (4 items). Participants rated their experience on a 7-point scale in response to each item ranging from 1 (maximum impairment) to 7 (no impairment). Individual items were equally weighted, and domain scores were calculated as the mean of all items within each domain; domain score range: 1 (maximum impairment) to 7 (no impairment). Participants with 0.5 point improvement from baseline in the domain scores were observed.
Time Frame: Day 393
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
percentage of participants
  Day 393: Dyspnea (n=42, 37) | 28.6 | 32.4
  Day 393: Fatigue (n=42, 37) | 35.7 | 35.1
  Day 393: Emotional function (n=42, 37) | 35.7 | 27.0
  Day 393: Mastery (n=42, 37) | 47.6 | 37.8

10. Secondary Outcome: Change From Baseline in Body Mass Index, Airflow Obstruction, Dyspnea, and Exercise Capacity (BODE) Scores at Day 393
Description: The BODE index is a multi-dimension COPD grading system that incorporates body-mass index (B), degree of airflow obstruction (O), dyspnea (D), and exercise capacity (E) as measured by the modified medical research council (MMRC) dyspnea scale and the 6-minute walk test. The MMRC dyspnea scale is a 5-point scale that measures the level of dyspnea (trouble breathing) experienced by participants where score range is 0 (none) to 4 (very severe ). BODE score is derived into a score range of 0 (healthy) to 10 (severe COPD).
Time Frame: Baseline, Day 393
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Benralizumab 100 mg
Number analyzed (Participants) | 42 | 40
units on scale
  Baseline (n=40, 39) | 2.8 (2.0) | 2.9 (1.8)
  Change at Day 393 (n=37, 32) | -0.1 (1.4) | -0.5 (1.4)

ADVERSE EVENTS:
Time Frame: Day 1 to 561
Arm/Group | Placebo | Benralizumab 100 mg
Serious Adverse Events (participants affected / at risk) | 9/50 | 14/51
Other Adverse Events (participants affected / at risk) | 41/50 | 44/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Benralizumab 100 mg (N=51)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (3) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (8)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Benralizumab 100 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 3 (3)
Injection site inflammation (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 5 (8)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (2)
Sinusitis (Infections and infestations) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Breath sounds abnormal (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (7)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 25 (62) | 26 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Aortic arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.